CLINICAL TRIAL: NCT03530735
Title: Finger-prick Autologous Blood (FAB) for Use in Dry Mouth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bedford Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 228680
Record Dates: First submitted 2018-04-10; First posted 2018-05-21 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-05

CONDITIONS: Xerostomia; Xerostomia Due to Radiotherapy; Xerostomia Due to Hyposecretion of Salivary Gland
Keywords: Fingerprick Autologous Blood
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fingerprick Autologous Blood (FAB) for Use in Dry Mouth (Experimental): All patients recruited will receive a 10ml saline mouth wash. Half will produce a blood-saline mixture from this mouthwash (preparation details below) and the other half will only use standard saline mouthwash. Each group will use their respective mouthwash 4 times a day for 4 weeks. During the following 4 weeks, participants will use the other mouthwash treatment. In the final 4 weeks, neither group of patients will be using either mouthwash.
  Patients will be assessed at week 0, 2, 4, 6, 8, 10 and 12. However only clinic visits 0, 4, 8 and 12 will require clinic visits. During weeks 2, 6, and 10 the patients will fill out the questionnaire at home.
  Interventions: Other: Finger-prick Autologous Blood (FAB)

INTERVENTIONS:
Other: Finger-prick Autologous Blood (FAB) — Patients will be instructed to use FAB therapy by:
  1. Hand hygiene with soap and water. Dry, then wipe their fingertip with an alcohol street before leaving to air dry.
  2. Use a diabetic lancet to prick their cleaned fingertip.
  3. Squeeze 5 drops of blood form their finger into 10ml of saline.
  4. Gargle the blood-saline mixture for 5 minutes.
  5. Swallow the blood-saline mixture.
  6. Repeat this 4 times per day.

SUMMARY:
This is a feasibility study that will assess the efficacy of using autologous blood to treat moderate to severe dry mouth. Dry mouth has been estimated to affect up to 64.8% of the general population (Navazesh et al., 2009) and many patients that are affected by Sjögren's syndrome or have had radiation therapy to combat head or neck cancer (Navazesh et al., 2009).

The blood will be applied to the interior of the mouth by means of a mouthwash. This research poses the first potential curative treatment for dry mouth - all other current dry mouth treatments are either symptomatic or lifestyle-based.

Autologous blood has been shown to be effective in treating the epithelial surface of dry eyes. This has been attributed to the analogous growth factors in the blood to that of tears - and potentially in this case, saliva - in healing the oral epithelial surface (Herbst et al., 2004).

DETAILED DESCRIPTION:
Fingerprick autologous blood (FAB) has been demonstrated to be effective in treating dry eye disease by inducing healing of the epithelial surface of the eye (Than et al., 2017). The epithelial layers of both the mouth and the eye require a non-vascular source of lubrication and nutrients (tears and saliva respectively). These nutrients include growth factors - naturally occurring substances capable of stimulating cellular growth. Saliva provides transforming growth factor alpha (TGF - α) (Mogi et al., 1995), epidermal growth factor (EGF) (Herbst, 2004; Marti et al., 1989), and Hepatocyte growth factor (HGF) (Amano et al., 1994) whilst tears provide EGF (Ohashi et al., 1989) amongst others (including TGF -β 1 and 2 (Gupta et al., 1996) integral to the proliferation, survival and differentiation of the oral epithelial cells (Klenkler et al., 2007). Therefore, as severe dry mouth disease (and a subsequent lack of saliva and growth factors) causes damage to the epithelial surface lining the mouth, a growth factor rich saliva substitute like FAB, should be an effective treatment for dry mouth. There is currently no study which details FAB for use in dry mouth.

Whole or parts of the three major salivary glands have been surgically transplanted or redirected to provide a replacement tear film in patients with severe dry eyes. This has been shown to be successful in both lubricating and improving eye comfort in afflicted patients (Geerling & Sieg, 2008). Since both blood and saliva have been shown to be effective as tear substitutes, it stands to reason that both tears and blood may be effective as a saliva substitute. Both tears and saliva are extraordinarily complex blood derived biological products which provide nourishment to an epithelial surface, and as such, blood should serve as a sufficiently close mimic of saliva.

Sjögren's syndrome, a chronic systemic autoimmune disease, occurs due to infiltration of secretory (exocrine) glands including the eye and mouth, resulting in dry eye and mouth respectively. FAB has been shown to be effective in treating Sjögren's induced dry eye and logically should also be an efficacious treatment for Sjögren's induced dry mouth.

Currently no curative measures for dry mouth exist. Oral dryness is managed conservatively by providing lubrication through a temporary solution such as lifestyle changes, artificial sprays, dry mouth mouthwash solutions or sialagogues (Shirlaw & Khan, 2017). There is no treatment that addresses the complexity of salivary constituents. Oral pilocarpine can be used to stimulate salivary glands at least as effectively as artificial saliva, however side effects were high including sweating, urinary frequency and vasodilation (Davies & Thompson, 2015).

Thus, FAB offers a potentially novel and better way than currently prescribed methods to treat dry mouth disease.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with dry mouth and are on or have refused treatment e.g. spray or mouthwash

Exclusion Criteria:

* Patients who do not have capacity to consent
* Patients with immunodeficiency
* Infected finger or systemic infection or on systemic antibiotics for infection
* Patients with active microbial infection, acute herpes simplex, herpes zoster or infected mouth ulcers
* Pregnant or breast feeding women
* Fear of needles and unwillingness to carry out repeated finger pricks
* Patients with frank oral ulceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of signs of clinical dry mouth | 6 months
  To assess improvement of signs of dry mouth using the Challachombe scale for visual identification and quantification of dry mouth
Improvement of symptoms of Dry Mouth | 6 months
  To assess improvement of signs of dry mouth using the seven item Xerostomia index.

SECONDARY OUTCOMES:
Adherence Self Report Questionnaire to assess patient compliance | 12 months
  We will create a questionnaire to assess patient adherence to apply fresh autologous blood during the study and after the study period has ceased. There will also be questions on patient comfort and thoughts on the application process.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navazesh M, Kumar SK. Xerostomia: prevalence, diagnosis, and management. Compend Contin Educ Dent. 2009 Jul-Aug;30(6):326-8, 331-2; quiz 333-4. PMID 19715009
- [Background] Herbst RS. Review of epidermal growth factor receptor biology. Int J Radiat Oncol Biol Phys. 2004;59(2 Suppl):21-6. doi: 10.1016/j.ijrobp.2003.11.041. PMID 15142631
- [Background] Than J, Balal S, Wawrzynski J, Nesaratnam N, Saleh GM, Moore J, Patel A, Shah S, Sharma B, Kumar B, Smith J, Sharma A. Fingerprick autologous blood: a novel treatment for dry eye syndrome. Eye (Lond). 2017 Dec;31(12):1655-1663. doi: 10.1038/eye.2017.118. Epub 2017 Jun 16. PMID 28622325
- [Background] Klenkler B, Sheardown H, Jones L. Growth factors in the tear film: role in tissue maintenance, wound healing, and ocular pathology. Ocul Surf. 2007 Jul;5(3):228-39. doi: 10.1016/s1542-0124(12)70613-4. PMID 17660896
- [Background] Mogi M, Inagaki H, Kojima K, Minami M, Harada M. Transforming growth factor-alpha in human submandibular gland and saliva. J Immunoassay. 1995 Nov;16(4):379-94. doi: 10.1080/15321819508013569. PMID 8567985
- [Background] Marti U, Burwen SJ, Jones AL. Biological effects of epidermal growth factor, with emphasis on the gastrointestinal tract and liver: an update. Hepatology. 1989 Jan;9(1):126-38. doi: 10.1002/hep.1840090122. PMID 2642290
- [Background] Amano O, Matsumoto K, Nakamura T, Iseki S. Expression and localization of hepatocyte growth factor in rat submandibular gland. Growth Factors. 1994;10(2):145-51. doi: 10.3109/08977199409010988. PMID 8068352
- [Background] Ohashi Y, Motokura M, Kinoshita Y, Mano T, Watanabe H, Kinoshita S, Manabe R, Oshiden K, Yanaihara C. Presence of epidermal growth factor in human tears. Invest Ophthalmol Vis Sci. 1989 Aug;30(8):1879-82. PMID 2788149
- [Background] Gupta A, Monroy D, Ji Z, Yoshino K, Huang A, Pflugfelder SC. Transforming growth factor beta-1 and beta-2 in human tear fluid. Curr Eye Res. 1996 Jun;15(6):605-14. doi: 10.3109/02713689609008900. PMID 8670763
- [Background] Geerling G, Sieg P. Transplantation of the major salivary glands. Dev Ophthalmol. 2008;41:255-268. doi: 10.1159/000131094. PMID 18453774
- [Background] Shirlaw PJ, Khan A. Oral dryness and Sjogren's: an update. Br Dent J. 2017 Nov 10;223(9):649-654. doi: 10.1038/sj.bdj.2017.882. PMID 29123309
- [Background] Davies AN, Thompson J. Parasympathomimetic drugs for the treatment of salivary gland dysfunction due to radiotherapy. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD003782. doi: 10.1002/14651858.CD003782.pub3. PMID 26436597